CLINICAL TRIAL: NCT06663761
Title: Correlation of Pain Intensity Measurements in Healthy Volunteers Exposed to Unpleasant Stimuli
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Radosław Owczuk, Prof., Medical University of Gdansk
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KB/259/2024
Record Dates: First submitted 2024-07-21; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Stimuli Responsive Polymers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental group (Experimental): Participants will be exposed to unpleasant stimuli, and their response will be determined.
  Interventions: Behavioral: Stimuli

INTERVENTIONS:
Behavioral: Stimuli — Stimuli (the order of stimuli 1-4 will be electronically randomized), with a break time between stimuli of 5-10 minutes:
  1. Non-invasive blood pressure measurement
  2. Heat
  3. Mechanical stimulation
  4. Visual stimulation
  5. Cold pressor test
  6. Spicy taste

SUMMARY:
Pain is an unpleasant sensory and emotional phenomenon that can be caused by tissue damage or potentially harmful stimuli. Pain is by definition a subjective phenomenon, and everyone experiences it differently, which creates problems in its assessment and treatment. There are many ways to measure pain, both through patient self-report (scales) and objective physiological indicators. However, there is no single, universal tool for measuring pain intensity that is simultaneously reliable, valid, and easy to use. Moreover, there are reports showing that not only the intensity of the unpleasant experience but also the nature of the stimulus can cause different levels of changes in the used indicators and scales. In this project, we will compare two devices used for pain monitoring based on physiological parameters: PainMonitor (Med-Storm, Oslo, Norway) and ANI Monitor (MetroDoloris, Loos, France). PainMonitor is a device that records skin conductance (SC) as an indicator of pain intensity. SC reflects the level of autonomic nervous system arousal. The device automatically analyzes these parameters and provides a numerical indicator of pain intensity/anesthesia level. The ANI Monitor is a device based on the analysis of parasympathetic nervous system activity through heart rate variability analysis. Based on this, the device also assesses the degree of pain intensity and presents it in numerical form. The aim of the project is to investigate the correlation between PainMonitor and ANI as tools for measuring pain intensity in situations where healthy volunteers are exposed to various unpleasant stimuli.

The study will involve approximately 100 healthy adult participants who will be exposed to three types of standardized stimuli: thermal (hot and cold), mechanical (pressure from a blood pressure cuff, pressure on a skin fold), chemical (spicy taste), and visual. Simultaneously, they will be monitored by PainMonitor, ANI, ECG, and peripheral perfusion index (using pulse oximetry). This data will then be compared and subjected to statistical analysis to determine if there is a relationship between the nature of the stimuli used and the objective and subjective indicators of pain intensity.

Stimuli (the order of stimuli 1-4 will be electronically randomized), with a break time between stimuli of 5-10 minutes:

1. NON-INVASIVE BLOOD PRESSURE MEASUREMENT: Non-invasive blood pressure measurement (NIBP) (single automatic blood pressure measurement using a Phillips IntelliVue Monitor).
2. HEAT: A metal cube with a temperature of 45 degrees Celsius will be used for heat stimulation. The cube will be applied for 60 seconds to the inner side of the forearm of the participant's dominant hand. The appropriate temperature of the cube will be maintained by keeping it in a water bath.
3. ALGOMETER: For mechanical stimulation, the researcher will apply pressure to the skin fold between the second and third fingers of the dominant hand using an algometer. The pressure will gradually increase from 0 to 250-300 kilo Pascal (kPa) and be maintained for 60 seconds.
4. VISUAL STIMULUS: For visual stimulation, a video will be shown on a display in front of the participant, depicting a model having a short intravenous cannula inserted. Participants will be asked to imagine that the hand on the screen is their own.
5. COLD: "Cold pressor test" - The participant's forearm will be immersed in water at a temperature of 2 degrees Celsius for 60 seconds or until discomfort causes the participant to withdraw their hand.
6. SPICY TASTE: 0.5 ml of spicy sauce with a specified amount of Scoville units will be applied to the participant's tongue using a syringe.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) general condition assessment 1 or 2
* age 18 - 40 yrs

Exclusion Criteria:

* any arrhythmia,
* taking medications from the groups of beta-blockers, gabapentinoids, benzodiazepines, painkillers within the last 12 hours,
* chronic pain conditions,
* pregnancy,
* trypanophobia (fear of needles)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain Monitor Measurements. | Continuously throughout whole study - approximately 1.5 hours
  Skin conductance will be recorded using PainMonitor (Med-Storm, Oslo, Norway) - on the non-dominant hand.
Heart rate and its variability (HRV) - high frequencies | Continuously throughout whole study - approximately 1.5 hours
  Heart rate and its variability (HRV) will be recorded using a Holter ECG monitor - electrodes on the chest. Frequency domain method will be used. The number of NN (beat to beat) intervals that match high frequency band (0.15 to 0.4 Hz) will be recorded.
Heart rate and its variability (HRV) - low frequencies | Continuously throughout whole study - approximately 1.5 hours
  Heart rate and its variability (HRV) will be recorded using a Holter ECG monitor - electrodes on the chest. Frequency domain method will be used. The number of NN (beat to beat) intervals that match low frequency band (0.04 to 0.15 Hz) will be recorded.
The analgesia-nociception index (ANI) | Continuously throughout whole study - approximately 1.5 hours
  The analgesia-nociception index (ANI) will be recorded using a dedicated device (MetroDoloris, Loos, France).
Perfusion index (PI) | Continuously throughout whole study - approximately 1.5 hours
  Perfusion index (PI) will be recorded using the pulse oximeter of the Phillips IntelliVue monitor - index finger of the non-dominant hand.
Subjective discomfort/pain - NRS | After each stimuli - approximately 1.5 hours
  Subjective discomfort/pain will be monitored using the Numerical Rating Scale (NRS, 0-10).
Subjective discomfort/pain - McGill Pain Questionnaire | After each stimuli - approximately 1.5 hours
  Subjective discomfort/pain will be monitored using the McGill Pain Questionnaire (SF-MPQ).

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Gdansk - Departament of Anesthesiology and Intensive Care, Gdansk, Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No